CLINICAL TRIAL: NCT07175506
Title: A Randomized, Double-blind, Placebo-controlled Phase I Clinical Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of CM559 in Healthy Subjects With Single Ascending Dose Administration
Brief Title: Study of CM559 in Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM559-109001
Record Dates: First submitted 2025-09-05; First posted 2025-09-16 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- CM559 or matched placebo cohort 1 (Experimental)
  Interventions: Drug: Placebo; Biological: CM559
- CM559 or matched placebo cohort 2 (Experimental)
  Interventions: Drug: Placebo; Biological: CM559
- CM559 or matched placebo cohort 3 (Experimental)
  Interventions: Drug: Placebo; Biological: CM559
- CM559 or matched placebo cohort 4 (Experimental)
  Interventions: Drug: Placebo; Biological: CM559
- CM559 or matched placebo cohort 5 (Experimental)
  Interventions: Drug: Placebo; Biological: CM559

INTERVENTIONS:
Drug: Placebo — Placebo injection administered IV, once.
Biological: CM559 — CM559 injection administered IV, once.

SUMMARY:
This study is a single center, randomized, double-blind, placebo-controlled, single dose, dose escalation Phase I clinical study aimed at evaluating the safety, tolerability, pharmacokinetics, pharmacodynamics, and immunogenicity of CM559 administered intravenously at different doses in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age ≥ 18 years & ≤60 years.
* Subjects voluntarily signed the Informed Consent Form and were able to comply with the provisions of this protocol.

Exclusion Criteria:

* The average number of cigarettes smoked per day is greater than 5 within 3 months prior to screening.
* Drinking heavily within 3 months prior to screening, or unable to guarantee not to drink alcohol during the research period, or positive alcohol breath testing.
* History of drug abuse within 1 year prior to screening, or positive urine drug abuse screening.
* Blood donation or any other form of blood loss exceeding 400mL, or accepting blood transfusion within 12 weeks prior to screening.
* Suspected allergy to Aβ-antibody drugs, humanized monoclonal antibody drugs and their excipients, or other biological agents, or have a history of severe allergic reactions to other drugs.
* Severe trauma or undergo major surgery within 3 months prior to screening,or planned surgery during the research period.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of single dose administration of CM559 in healthy male subjects: Adverse events (AEs), physical examinations, vital signs, 12-lead electrocardiograms (ECGs), magnetic resonance imaging (MRI), laboratory tests, etc. | Up to 99 Days
  All adverse events (AEs) collected from all subjects from the time of signing the informed consent form (ICF) to the completion of the study (or early withdrawal), including clinical manifestations, severity, occurrence time, end time, treatment measures, and outcomes, as well as their correlation with the investigational drug.
  Any clinically significant abnormalities found during the physical examinations, vital signs examination, ECGs examinations and laboratory tests.
  The proportion of subjects experienced amyloid-related imaging abnormalities (ARIA) identified by MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Mengchang Yang, Study Chair — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China